CLINICAL TRIAL: NCT03617718
Title: Methods to Identify and Treat Severe Asthma Patients Project 2: Airway pH Phenotyping
Brief Title: Project 2 Airway Potential Hydrogen (pH) in Asthma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Kristie Ross, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-18-28; P01HL158507 (NIH)
Record Dates: First submitted 2018-07-19; First posted 2018-08-06 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis; Asthma; Severe Persistent Asthma; Healthy
MeSH Terms: conditions — Cystic Fibrosis; Asthma

STUDY DESIGN:
Intervention Model Description: All participants will go through the same study procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cystic Fibrosis (Experimental): All Cystic Fibrosis participants will undergo screening, baseline characterization, a non-invasive challenge test with inhaled alkaline glycine buffer, followed by repeated measurements of airway function and inflammation, and a research bronchoscopy.
  Interventions: Drug: Glycine Buffer
- Asthma (Experimental): All Asthma participants will undergo screening, baseline characterization, a non-invasive challenge test with inhaled alkaline glycine buffer, followed by repeated measurements of airway function and inflammation, and a research bronchoscopy.
  Interventions: Drug: Glycine Buffer
- Healthy Control (Experimental): All Healthy Control participants will undergo screening, baseline characterization, a non-invasive challenge test with inhaled alkaline glycine buffer, followed by repeated measurements of airway function and inflammation, and a research bronchoscopy.
  Interventions: Drug: Glycine Buffer

INTERVENTIONS:
Drug: Glycine Buffer — Subjects will be asked to perform an Inhaled Glycine Buffer followed by a series of Pulmonary Function Tests (PFTs) and then a research bronchoscopy will happen at visit 3.

SUMMARY:
This study is testing a non invasive way to measure airway pH in individuals with Asthma and Cystic Fibrosis using a new inhaled drug. The airway pH will help health care providers in creating tailored treatment plans for individuals suffering from these specific conditions.

DETAILED DESCRIPTION:
Asthma can affect patients in different ways. Some of the differences in how severe asthma is or how well patients respond to asthma medicines are due to differences in the biology of the airways or breathing tubes. The pH of the airway, which is a measure of the balance between acids and bases in our airways, is one example of how differences in biology can affect asthma and other lung diseases. Airway pH can be measured during a procedure called a bronchoscopy, in which a camera is inserted into the airways or breathing tubes. The lower the pH, the more acid is present. People with lower airway pHs, or more acid present in their airways/breathing tubes, tend to have more trouble with their asthma.

The pH value or acid level in the airway plays a role in respiratory function (breathing) and preventing inflammation (swelling) in the respiratory tract (throat, airways, and lungs). Studies have found that in individuals with asthma, Cystic Fibrosis (CF) and other pulmonary disorders, a lower pH value is present in the airway when compared to healthy individuals. Studies have also found that patients with asthma have a lower airway pH during asthma flares, and may affect how well some breathing medicines work. If we can better identify the changes in the airways or breathing pipes in patients with asthma and CF, we may be able to help patients make better choices about the medicines or treatments that are most likely to work best for each patient.

Right now the only way to measure airway pH is with a bronchoscopy procedure. During a bronchoscopy, a scope with a camera is inserted into the breathing tubes, often under sedation in a special procedure area. This research study is being done to test if we can measure how acidic the airway is in a simple and non-invasive test that can be done in a doctor's office.

This non-invasive diagnostic test, called a Glycine Buffer Challenge test, may be able to identify which asthma and CF patients have low airway pH levels. We are also studying the phenotypes (observable traits) in asthma and CF patients with decreased airway pH values. If this research study is successful, in the future (after this research study is done) we may be able to offer better ways to treat patients with low airway pH.

The Glycine Buffer Challenge test includes giving an investigational drug to breathe in (inhale). The investigational drug is the Glycine Buffer. "Investigational" means the drug is not approved by any regulatory agencies including the Food and Drug Administration (FDA), and is still being tested for safety and effectiveness. The research is registered with the FDA, but again the Glycine Buffer treatment in this study administered (during the Glycine Buffer challenge testing) is not an approved treatment or diagnostic test for asthma.

The study will enroll a total of 75 volunteers; 50 volunteers with severe asthma, 15 volunteers with cystic fibrosis, and 10 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Subjects with Severe Asthma

1. Asthma diagnosis established during at least 3 months of evaluation and care by an asthma specialist (pulmonologist or allergist).
2. Adult male or female age ≥ 18 and ≤ 50 years at the time of enrollment
3. Forced expiratory volume in 1 second (FEV1) bronchodilator reversibility > 12% or methacholine FEV1 by 20% of baseline (PC20) < 16 mg/ml (historical methacholine data from previous NIH trial including Severe Asthma Research Program (SARP) or Asthma Network (AsthmaNet) will be allowed).
4. If FEV1 is <50% predicted, precluding methacholine challenge testing, investigator acceptance of the diagnosis of asthma is acceptable
5. Treatment with high-dose inhaled corticosteroids (> 880 mcg fluticasone or highest marketed equivalent/day) along with a second controller or systemic corticosteroids for at least 3 months prior to enrollment and for at least 6 of the last 12 months.
6. Lack of asthma control despite this treatment evidenced by any one of the following:

   1. Asthma Control Questionnaire (ACQ) > 1.5 or Asthma Control Test (ACT) < 20
   2. >2 bursts of systemic corticosteroids (3 days or more) in the previous 12 months
   3. >1 hospitalization or ICU stay for acute asthma in the previous 12 months
   4. Mild to moderate obstructive lung disease with 45%< FEV1 < 80% predicted (with low FEV1/FVC) prior to bronchodilator
7. Post bronchodilator FEV1 < 55% predicted on the day of study procedures including the Inhaled glycine buffer challenge test and bronchoscopy. (These events may be rescheduled in the event participants meet all inclusion criteria at the time of screening)

Healthy Volunteers

1. Adult males or females age ≥ 18 and ≤ 50 years at time of enrollment
2. Non-smokers
3. No history of asthma, chronic obstructive pulmonary disease (COPD), or other chronic lung disease
4. No history of severe allergic/atopic disease requiring immunotherapy or immunomodulators

Subjects with Cystic Fibrosis

1. Adult male or female age ≥ 18 and ≤ 50 at time of enrollment
2. Confirmed diagnosis of CF as evidenced by 1 or more clinical features consistent with the CF phenotype and 1 or more of the following laboratory criteria:

   1. Sweat chloride equal to or greater than 60 m/Eq/L by quantitative pilocarpine iontophoresis test (Sweat Test)
   2. Two well-characterized disease causing mutations in the Cystic fibrosis transmembrane conductance regulator (CFTR) gene.
3. Weight > 50 kg at screening visit
4. Mild obstructive lung disease defined as post bronchodilator baseline FEV1 > 70% predicted for age, height and gender
5. Clinically stable with no significant changes in health status within 4 weeks, including FEV1 within 10% of baseline, at the time of screening (may be rescreened)

Exclusion Criteria:

General (applying to all participants)

1. > 5 pack year smoking history
2. Body mass index (BMI) greater than 45
3. Unable to perform repeatable consistent efforts in pulmonary function testing
4. Individuals with prior diagnosis of vocal cord dysfunction or an anatomic anomaly that would increase the risks associated with the bronchoscopy procedure
5. Prior diagnosis of any chronic lung disease that in the investigator's opinion would make them unsuitable for study participation
6. History of premature birth before 35 weeks gestation
7. Planning to relocate away from the clinical center (Cleveland, Ohio) area before study completion
8. Lack of reliable communications channel (hard-wire phone, cell phone, email for follow-up contacts after bronchoscopy)
9. Allergic to anesthetic medication(s) that would prevent participation in the study's bronchoscopy
10. Blood pressure parameters outside the normal range of 90-180 mm Hg systolic and 50-100 mm Hg diastolic at time of screening
11. Individuals with diabetes mellitus (type 1 or type 2) (subjects with CF who have CF related diabetes may be enrolled)
12. Individuals with renal failure or creatinine > 1.8 mg/dl at time of screening
13. Individuals who are pregnant, breastfeeding, or are unwilling to use a medically acceptable method of birth control (as indicated on the Birth Control Methods Reference Card) from the time of consent until the end of the study to avoid pregnancy
14. Individuals who report additional chronic diseases requiring medication of the heart, lungs, kidney, liver, brain, etc., or afflicted with any acute or chronic pathology that in the opinion of the screening physician makes them unsuitable for study such as coronary artery disease
15. Respiratory or other infection requiring systemic antibiotics within the previous 14 days (can be rescreened)
16. Current use of a vitamin K antagonist (warfarin) or other anticoagulant (e.g., heparin, clopidogrel, enoxaparin or dalteparin)
17. Current use of beta-adrenergic blockers, tricyclic antidepressants, meperidine (or related central nervous system (CNS) agents), or nitrates
18. Inherited or acquired blood coagulation disorder, congenital methemoglobinemia, or a familial hemoglobinopathy that impacts oxygen delivery (e.g., sickle cell)
19. Any illness, condition or recent surgeries that may increase the risks associated with the study
20. Participation in an investigational drug study within the 4 week period prior to screening (Visit 1)

Severe Asthma specific exclusion criteria

1. Asthma exacerbation within 4 weeks prior to screening (Visit 1) (may be rescreened)
2. Initiation of new chronic treatment or change in dose of chronic treatment for asthma within 2 months of screening
3. Intubation for asthma within the past 12 months
4. More than 3 exacerbations within the past 6 months

Cystic fibrosis specific exclusion criteria

1. Positive sputum culture for Burkholderia cepacia complex organism within the previous 12 months
2. Active treatment for non-tuberculous mycobacterium
3. International Normalized Ratio (INR) > 1.2 at time of screening
4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 times the upper limit of normal at screening, history of biliary cirrhosis or portal hypertension
5. Treatment with Kalydeco (ivacaftor) within 12 weeks of screening
6. History of pulmonary hypertension
7. Severe malnutrition
8. Pulse oximetry < 92% at screening or chronic use of supplemental oxygen
9. Currently listed for lung or other organ transplantation
10. Pneumothorax within 2 years
11. Hemoptysis other than trace during the past 12 months or history of life threatening hemoptysis ever
12. Initiation of any new chronic treatment with 4 weeks of screening (can be rescreened)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Changes in Fractional Exhaled Nitric Oxide (FeNO) levels | Baseline, every 15 minutes after administration of glycine buffer for 60 minutes
  FeNO measurements will be compared among the three different participant groups (Cystic Fibrosis, Severa Asthma and Healthy Volunteers).
Frequency of shared phenotypic features among participants with low airway pH compared to those with low exhaled breath condensate (EBC) pH | Baseline, 3 months
  The number of times that the phenotypic features of low EBC pH ( high BMI (>30), low methacholine PC20 (<5), age, and bronchoalveolar lavage neutrophils) are also shared with participants that are found to have a low airway pH.
Large airway pH as measured by bronchoscopy | Visit 3 (day 21)
Middle airway pH as measured by bronchoscopy | Visit 3 (day 21)
Lower airway pH as measured by bronchoscopy | Visit 3 (day 21)

CONTACTS AND LOCATIONS:
Overall Officials: Kristie R Ross, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (2):
- United States (2):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University Hospitals Cleveland Medical Center - Asthma Research Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification and analysis will be shared.
Supporting Information: SAP, CSR
Time Frame: Available Immediately following publication. No end date
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.